CLINICAL TRIAL: NCT02794194
Title: Effects of a Whole Body Vibration Training on Unstable Surface in Recreational Athletes With Chronic Ankle Instability
Brief Title: Effects of Whole Body Vibration Training on Unstable Surface
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LRRD2016/001
Record Dates: First submitted 2016-05-27; First posted 2016-06-09 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Ankle Instability
Keywords: Chronic Ankle Instability; Whole Body Vibration; Proprioception

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (3):
- Control group (No Intervention): No intervention
- Vibration group (Experimental): Proprioceptive training on a whole body vibration platform. Participants in the Vibration group trained with a BOSU® on a Fitvibe Excel Pro vibration platform (Fitvibe, Bilzen, Belgium).
  Interventions: Other: Proprioceptive training on a whole body vibration platform
- Non-vibration group (Experimental): Proprioceptive training with the BOSU® on the floor. Participants in the Non-Vibration group trained with a BOSU® on the floor.
  Interventions: Other: Proprioceptive training with the BOSU® on the floor

INTERVENTIONS:
Other: Proprioceptive training on a whole body vibration platform — The Training programme consisted of three series of 4 exercises of 45 seconds with 45 seconds rest between exercises. In this intervention participants trained with the BOSU® on a Fitvibe Excel Pro vibration platform (Fitvibe, Bilzen, Belgium).
  Arms: Vibration group
Other: Proprioceptive training with the BOSU® on the floor — The Training programme consisted of three series of 4 exercises of 45 seconds with 45 seconds rest between exercises. In this intervention participants trained with the BOSU® on the floor.
  Arms: Non-vibration group

SUMMARY:
After an initial ankle sprain, Chronic Ankle Instability is one of the most common residual symptoms which include pain, swelling, recurrent sprain, episodes of ankle joint "giving away" or decreased function. Recently, Whole Body Vibration (WBV) training has been introduced as a preventive and rehabilitative tool. It can be hypothesized that WBV on unstable surfaces might enhance neuromuscular control. Therefore, the aim of this study was to investigate the effects of a 6-week WBV training on an unstable surface on body composition, balance, strength and reflex and muscle activity of ankle muscles in recreational athletes with CAI.

DETAILED DESCRIPTION:
Participants:

Fifty physically active recreational athletes with self-reported CAI volunteered to participate in the study. These subjects were assigned to one of three groups: the Vibration group (VIB), Non-Vibration group (N-VIB) and Control group (CON).

Each participant was informed of the risks and discomforts associated with this investigation and signed an informed consent document before the onset of the experiments. The experimental protocol was approved by the Ethics Committee of Clinical Research at the Hospital Complex in Toledo (Spain).

Procedures:

The investigators performed a randomized clinical trial with a cross over design. Participants were assessed at three time points: pre-training (Pre), post-training 1 (Post1) and post-training 2 (Post2) (6 weeks after the last training session). Measurements consisted in a body composition analysis, two balance tests, a forced ankle inversion test and an isokinetic strength test. Assessors and the researcher who performed the statistical analysis were blinded to group allocation. Measurements and the training protocol were developed in the Performance and Sport Rehabilitation Laboratory at the University of Castilla-La Mancha (Toledo, Spain).

Training protocol:

Participants followed a balance training protocol of six weeks for an unstable ankle. Exercises sessions were performed three days a week (48 hours between sessions) on a BOSU® Balance Trainer. All the exercises were carried out only on the unstable ankle and were the same for both experimental groups. Participants in the N-VIB group trained with the BOSU® on the floor, whereas participants in the VIB group trained with the BOSU® on a Fitvibe Excel Pro vibration platform (Fitvibe, Bilzen, Belgium). The Training programme consisted of three series of 4 exercises of 45 seconds with 45 seconds rest between exercises. Following the recommendations of a previous research study18, the level of difficulty was increased in all exercises after three weeks. Also, frequency was progressively increased every two weeks.

Biodex Balance System test:

Ankle balance was assessed with the Biodex Stability System (Biodex Medical Systems, Shirley, New York, USA). The balance test consist of a mobile platform, which allows up to 20° of surface tilt in a 360° range of motion. The platform, which interfaced with computer software (Biodex, Version 1.32, Biodex Medical System), generates three stability indexes: Overall, which represents the platform displacement in all directions; Anterior/Posterior and Medial/Lateral.

The test was performed at level 8 with participants barefoot at single-leg stance. Participants were asked to step on the platform with eyes open and assume a comfortable position while maintaining slight flexion in the knees (15°), to look straight ahead at the monitor and to place their hands in their hips. Foot position coordinates were registered to ensure the same position was used in all tests.

Star Excursion Balance Test (SEBT):

The SEBT, was performed with the participants standing barefoot in the middle of a grid formed by eight tape measures extending out at 45° from each other, each of which was labelled according to the direction of excursion in relation to the standing leg. Participants were asked to maintain a single-stance while reaching with the contralateral leg to touch lightly as far as possible along the chosen direction with the most distal part of their foot and then return to bilateral stance. A standardised protocol of 4 practice trials followed by 3 test trials was performed in each of the eight directions to minimize the learning effect. Reach distances were measured by the same researcher making a mark on the tape measure. The average of the three test trials normalised to leg length of the stance leg was used for analysis.

Body composition:

Height was measured using a wall-mounted stadiometer (model 220, Seca, Hamburg, Germany). Body weight (in underwear) was measured with a digital balance (model 707, Seca, Hamburg, Germany; weighing accuracy of 0.1 kg). Total and regional body composition was measured by dual energy X-ray absorptiometry (Lunar iDXA; GE-Healthcare, Fairfield, CT, USA) using a standardized protocol specified by the manufacturer. Lean mass, fat mass, %fat, bone mineral content and bone mineral density for the total body and for the leg with ankle instability were obtained using the enCORE software (GE Healthcare, v. 13.40).

Inversion test:

Electromyographic (EMG) measurements were taken from the peroneus longus (PL), peroneus brevis (PB) and tibialis anterior (TA). The test was performed on a custom-designed ankle inversion platform capable of producing a 30⁰ inversion, previously used in other research. The start and the end of the inversion was marked by a double axis goniometer (SG110/A, Biometrics Ltd, Gwent, UK) attached to the platform doors to detect any change in the angle of the doors.

Muscular activity was recorded using a portable eight channel telemetry and data logger (ME6000-T8, Mega Electronics, Kuopio, Finland) and was analysed using MegaWin 3.1-b10 software (Mega Electronics, Kuopio, Finland).

Isokinetic test:

Ankle evertor muscles were tested on a Biodex Multi-Joint System 3 dynamometer (Biodex Medical System, New York, USA) at three different velocities: 60, 180 and 300 degrees per second for eccentric and concentric contractions. The isokinetic test was carried out on two different days. The first day, participants were familiarized with the testing procedure and the position on the dynamometer for each participant was registered to ensure that the test was carried out always under the same conditions. Measurements were taken on the second day.

Data analysis:

Statistical analysis was performed using IBM SPSS Statistics v.22.0 (SPSS Inc., Chicago, Illinois, USA). The level of significance was set at p < 0.05. The normality of each variable was initially tested with the Shapiro-Wilk test. All the variables presented a normal distribution. A 2-way repeated measures analysis of variance (ANOVA) was performed for all outcome variables to analyze the interaction between groups (VIB, N-VIB, CON) and the time of assessment (pre-training, post-training 1, post-training 2). The Bonferroni multiple comparison test was performed to account for multiple comparisons. The effect size was calculated in all pairwise comparisons. The magnitude of the effect size was interpreted using Cohen's scale. All the data were presented as mean and standard deviation.

ELIGIBILITY:
Inclusion Criteria:

* History of at least 1 significant ankle sprain (the most recent injury must have occurred more than 3 months prior to study enrolment).
* 2 or more episodes of the ankle giving way in the last 6 months.
* A score of ≤24 on the Spanish version of the Cumberland Ankle Instability Tool.
* Age range: 18-30 years.

Exclusion Criteria:

* History of previous surgeries to the musculoskeletal structures in either lower extremity.
* History of a fracture in either lower extremity requiring realignment.
* An acute injury to musculoskeletal structures of other joints of the lower extremity in the previous 3 months that impacted joint integrity and function, resulting in at least 1 interrupted day of desired physical activity.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in electromyographic activity | baseline, after the completion of the intervention, and 6 weeks after the completion of the intervention
  Baseline: before the initiation of the exercise programs (at most 7 days before the initiation of the exercise programs). First follow-up measurement: after the completion of the exercise programs (at most 7 days after the completion of the last training session. Average time period: six weeks after the initiation of the intervention). Second follow-up measurement: 6 weeks after the completion of the exercise programs (average time period: twelve weeks after the initiation of the intervention)
Change in muscle strength | baseline, after the completion of the intervention, and 6 weeks after the completion of the intervention
  Baseline: before the initiation of the exercise programs (at most 7 days before the initiation of the exercise programs). First follow-up measurement: after the completion of the exercise programs (at most 7 days after the completion of the last training session. Average time period: six weeks after the initiation of the intervention). Second follow-up measurement: 6 weeks after the completion of the exercise programs (average time period: twelve weeks after the initiation of the intervention)
Change in balance (Biodex Balance System test) | baseline, after the completion of the intervention, and 6 weeks after the completion of the intervention
  Baseline: before the initiation of the exercise programs (at most 7 days before the initiation of the exercise programs). First follow-up measurement: after the completion of the exercise programs (at most 7 days after the completion of the last training session. Average time period: six weeks after the initiation of the intervention). Second follow-up measurement: 6 weeks after the completion of the exercise programs (average time period: twelve weeks after the initiation of the intervention)
Change in balance (Star Excursion Balance Test (SEBT) | baseline, after the completion of the intervention, and 6 weeks after the completion of the intervention
  Baseline: before the initiation of the exercise programs (at most 7 days before the initiation of the exercise programs). First follow-up measurement: after the completion of the exercise programs (at most 7 days after the completion of the last training session. Average time period: six weeks after the initiation of the intervention). Second follow-up measurement: 6 weeks after the completion of the exercise programs (average time period: twelve weeks after the initiation of the intervention)

SECONDARY OUTCOMES:
Change in lean mass and fat mass (obtained using the enCORE software (GE Healthcare, v. 13.40) | baseline, after the completion of the intervention, and 6 weeks after the completion of the intervention
  Baseline: before the initiation of the exercise programs (at most 7 days before the initiation of the exercise programs). First follow-up measurement: after the completion of the exercise programs (at most 7 days after the completion of the last training session. Average time period: six weeks after the initiation of the intervention). Second follow-up measurement: 6 weeks after the completion of the exercise programs (average time period: twelve weeks after the initiation of the intervention)
Change in bone mineral content and bone mineral density (obtained using the enCORE software (GE Healthcare, v. 13.40) | baseline, after the completion of the intervention, and 6 weeks after the completion of the intervention
  Baseline: before the initiation of the exercise programs (at most 7 days before the initiation of the exercise programs). First follow-up measurement: after the completion of the exercise programs (at most 7 days after the completion of the last training session. Average time period: six weeks after the initiation of the intervention). Second follow-up measurement: 6 weeks after the completion of the exercise programs (average time period: twelve weeks after the initiation of the intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- Performance and Sport Rehabilitation Laboratory, Toledo, Toledo, Spain

REFERENCES:
- [Derived] Sierra-Guzman R, Jimenez JF, Ramirez C, Esteban P, Abian-Vicen J. Effects of Synchronous Whole Body Vibration Training on a Soft, Unstable Surface in Athletes with Chronic Ankle Instability. Int J Sports Med. 2017 Jun;38(6):447-455. doi: 10.1055/s-0043-102571. Epub 2017 May 9. PMID 28486729